CLINICAL TRIAL: NCT00848094
Title: Phase I Trial of Radiation Dose Escalation for Locally Advanced Hepatocellular Carcinoma
Brief Title: Radiation Dose Escalation Study for Advanced Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Guoliang Jiang, Fudan University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCR-003
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; radiation therapy; 3-dimensional conformal radiation therapy (3-DCRT); intensity modulated radiation therapy (IMRT); active breathing control
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1 (Other): Arm I: tumor diameter more than 5 cm and less than 10 cm.
  Interventions: Radiation: 3DCRT/IMRT
- arm 2 (Other): Arm II: tumor diameter no less than 10 cm.
  Interventions: Radiation: 3DCRT/IMRT

INTERVENTIONS:
Radiation: 3DCRT/IMRT — The starting radiation doses were the total tumor doses of 46 Gy in 2 Gy per fractions for arm I . Escalation was achieved by increasing the tumor dose of each cohort in increments of 4.0 Gy. Subsequent cohorts received higher doses up to a chosen maximum of 62 Gy for arm I.
  Arms: arm 1
Radiation: 3DCRT/IMRT — The starting radiation doses were the total tumor doses of 40 Gy in 2 Gy per fractions for arm II. Escalation was achieved by increasing the tumor dose of each cohort in increments of 4.0 Gy. Subsequent cohorts received higher doses up to a chosen maximum of 52 Gy for arm II.
  Arms: arm 2

SUMMARY:
The purpose of this clinical study is to determine the maximum tolerated dose (MTD) of 3-dimensional conformal radiation therapy (3-DCRT)/intensity modulated radiation therapy (IMRT) for locally advanced hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed or clinically diagnosed HCC
* Surgically unsectable or medically inoperable diseases, or surgery declined by the patient
* Solitary intrahepatic lesion with diameter bigger than 5 cm, without extrahepatic and/or distant metastases
* Associated with cirrhosis of Child-Pugh A
* Karnofsky performance status (KPS) of ≥ 70
* Normal renal function and adequate bone marrow reservation
* Tolerate active breathing control (ABC)

Exclusion Criteria:

* Child-Pugh B or C liver cirrhosis score
* Previous radiotherapy to the liver
* Indistinct tumor boundary in CT/MRI image

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Toxicity was graded using the CTCAE 3.0. Dose-limiting toxicity was defined as acute ≥ grade 3 hepatic or gastrointestinal toxicity, or any grade 5 treatment-related adverse event, or late complication of radiation-induced liver disease. | 4 months

SECONDARY OUTCOMES:
1,2 and 3 years survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Jiang, M.D., Principal Investigator — Fudan University